CLINICAL TRIAL: NCT04945577
Title: The Relationship Between Vitamin D Levels, Inflammatory Parameters and Disease Severity of COVID-19 Infection: A Retrospective Study
Brief Title: The Relationship Between Vitamin D Levels, Inflammatory Parameters and Disease Severity of COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Gulcanozturk
Record Dates: First submitted 2021-06-06; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Vitamin D Deficiency; Covid19
Keywords: COVID-19; Vitamin D; Disease severity; Inflammatory markers
MeSH Terms: conditions — Vitamin D Deficiency; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental: Mild Clinical Group: patients showing mild clinical symptoms without pneumonia.
  Interventions: Diagnostic Test: Inflammatory Parameters; Other: 25 OH Vitamin D Level
- Experimental: Moderate Clinical Group: patients with fever, other respiratory symptoms, and pneumonia findings based on radiological imaging
  Interventions: Diagnostic Test: Inflammatory Parameters; Other: 25 OH Vitamin D Level
- Experimental: severe/critical clinical group: severe one of these as follows; patients with hypoxia (≤93% oxygen saturation), respiratory distress (RR >30 times per minute), partial pressure of arterial blood oxygen (PaO 2 )/the fraction of inspired oxygen (FiO 2 ) ≤ 300 mmHg, patients whose chest imaging shows that lung damage develops significantly within 24 to 48 hours, or critical one of these as follows; respiratory failure requiring mechanical ventilation, signs of septic shock with multiple organ failure requiring intensive care unit admission.
  Interventions: Diagnostic Test: Inflammatory Parameters; Other: 25 OH Vitamin D Level

INTERVENTIONS:
Diagnostic Test: Inflammatory Parameters — Laboratory measurement of patient's inflammatory status in unit of % and mg/dl
Other: 25 OH Vitamin D Level — Laboratory measurement of patient's 25 OH vitamin D level in unit of ng/dl

SUMMARY:
Vitamin D deficiency increases the susceptibility to respiratory virus infections and the severity of infections. Inflammation plays a key role in pathogenesis in COVID19 while identifying clinical course and prognosis COVID19.The aim of this study was to determine the relationship between 25OH vitamin D levels, inflammatory laboratory parameters of neutrophil to lymphocyte ratio (NLR), platelet to lymphocyte ratio (PLR), C-reactive protein (CRP) levels and disease severity of COVID19 infection.

DETAILED DESCRIPTION:
In this retrospective study 300 patients diagnosed with COVID19 were included. According to clinical classification of cases with COVID19 the patients were divided into three groups; mild (Group1), moderate (Group2) and severe/critical (Group3). The 25OH vitamin D values below 20 ng/ml were defined as deficiency, 21-29 ng/ml were defined as insufficiency, and 30 ng/ml and above were defined as normal. Patients' age, gender, comorbid diseases and laboratory values were recorded

ELIGIBILITY:
Inclusion Criteria:

* The study included 300 polymerase chain reaction (PCR) test positive patients and whose 25-OH vitamin D levels were measured in the last 6 months

Exclusion Criteria:

* Patients with COVID-19 whose 25-OH vitamin D levels were not measured in the last 6 months before the COVID-19 diagnosis were excluded from the study

Ages: 16 Years to 97 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: COVID19 infection positive patients whose polymerase chain reaction (PCR) test positive patients and whose 25-OH vitamin D levels were measured in the last 6 months
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
25-OH vitamin D | 1 day
  laboratory measurement in unit of ng/ml
White blood cell count | 1 day
  laboratory measurement in unit of x103/uL
neutrophil count | 1 day
  laboratory measurement in unit of x103/uL
neutrophil ratio | 1 day
  laboratory measurement in unit of %
lymphocyte count | 1 day
  x103/uL
lymphocyte ratio | 1 day
  laboratory measurement in unit of %
platelet count | 1 day
  laboratory measurement in unit of x103/uL
hemoglobin count | 1 day
  laboratory measurement in unit of g/dl
C-reactive protein levels | 1 day
  laboratory measurement in unit of mg/dL
neutrophil to lymphocyte ratio | 1 day
  laboratory measurement in unit of %
platelet to lymphocyte ratio | 1 day
  laboratory measurement in unit of %

CONTACTS AND LOCATIONS:
Locations (1):
- Gulcan Ozturk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ali N. Elevated level of C-reactive protein may be an early marker to predict risk for severity of COVID-19. J Med Virol. 2020 Nov;92(11):2409-2411. doi: 10.1002/jmv.26097. Epub 2020 Jun 9. No abstract available. PMID 32516845
- [Background] Ali N. Role of vitamin D in preventing of COVID-19 infection, progression and severity. J Infect Public Health. 2020 Oct;13(10):1373-1380. doi: 10.1016/j.jiph.2020.06.021. Epub 2020 Jun 20. PMID 32605780
- [Background] Khemka A, Suri A, Singh NK, Bansal SK. Role of Vitamin D Supplementation in Prevention and Treatment of COVID-19. Indian J Clin Biochem. 2020 Oct;35(4):502-503. doi: 10.1007/s12291-020-00908-3. Epub 2020 Jul 30. No abstract available. PMID 32837034